CLINICAL TRIAL: NCT01533402
Title: Internet-delivered Cognitive Behavior Therapy (CBT) Treatment for Anxiety Disorders in Children Age 8-12 Years - a Randomised Controlled Trial
Brief Title: Internet-delivered Cognitive Behavior Therapy (CBT) for Children Age 8-12 Years With Anxiety Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); Barn-och ungdomspsykiatrin (BUP), Stockholm (Unknown)
Responsible Party: Principal Investigator, Eva Serlachius, Principal Investigator, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/2027-31/5
Record Dates: First submitted 2012-02-06; First posted 2012-02-15 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Anxiety Disorders
Keywords: Cognitive behavior therapy; Internet; Anxiety disorders; Children
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attention control (Placebo Comparator): Weekly support from therapist without CBT-interventions
  Interventions: Behavioral: therapist support
- Internet CBT (Experimental): Internet-delivered cognitive behavioural therapy with therapy support
  Interventions: Behavioral: Internet-delivered CBT

INTERVENTIONS:
Behavioral: therapist support — Weekly therapist support without CBT-interventions
  Arms: Attention control
Behavioral: Internet-delivered CBT — Internet-delivered cognitive behavioural therapy with therapist support
  Arms: Internet CBT

SUMMARY:
The purpose of this study is to investigate whether a 10 week Internet-delivered CBT is a feasible approach to treat children (age 8-12 years) with anxiety disorder (social phobia, panic disorder, specific phobia, generalized anxiety disorder or separation anxiety disorder). The program is directed toward both the parents and children. The patients work with the treatment is supported through on-line contact with a therapist. Approximately 128 patients will be included in the study and randomized to either condition. All included patients are assessed before the treatment starts and after 10 weeks (post treatment). Follow-up assessments are conducted at 3 and 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of social phobia, panic disorder, specific phobia, generalized anxiety disorder or separation anxiety disorder,
* age between 8 and 12 years,
* ability to read and write Swedish and
* with access to a computer and use of internet.

Exclusion Criteria:

* Presence of neuropsychiatric diagnosis or a primary psychiatric disorder other than those that the treatment aims at.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Anxiety symptoms | two - three weeks pre treatment and 10 weeks, 3 months and 12 months post treatment
  Change from baseline in anxiety symptoms. Clinician Severity Rating (CSR) assessed by a clinician with Anxiety Diagnostic Interview Schedule (ADIS C/P).

SECONDARY OUTCOMES:
Anxiety symptoms | two weeks pre treatment and 10 weeks, 3 months and 12 months post treatment
  Change from baseline in anxiety symptoms. Fear Survey Schedule for Children (FSSC-C/P).
Quality of Life | two weeks pre treatment and 10 weeks, 3 months and 12 months post treatment
  Quality of Life (QOLI)
comorbidity | two - four weeks before treatment starts
  Development and Wellbeing Assessment (DAWBA)
Depressive symptoms | two weeks pre treatment and 10 weeks, 3 months and 12 months post treatment
  Children Depression Scale (CDI)
Funtional impairment | two weeks pre treatment and 10 weeks, 3 months and 12 months post treatment
  Children´s Global Assessment Scale (CGAS)
Client Satisfaction Scale | two weeks before treatment and 10 weeks, 3 and 12 months post treatment
  Client Satisfaction Scale (CSS)
Parental psychopathology | two weeks pre treatment
  Primary Care Evaluation of Mental disorders (Prime-MD)
Anxiety symptoms | two weeks pre treatment and 10 weeks, 3 months and 12 months post treatment
  Change from baseline in anxiety symptoms. Penn State Worry Questionnaire for Children (PSWQ-C).
Anxiety symptoms | two weeks pre treatment and 10 weeks, 3 months and 12 months post treatment
  Change from baseline in anxiety symptoms. Separation Anxiety Inventory for Children (SAI-C/P)
Anxiety symptoms | two weeks pre treatment and 10 weeks, 3 months and 12 months post treatment
  Change from baseline in anxiety symptoms. Social Phobia and Anxiety Inventory (SPAI-C/P)
Anxiety symptoms | two weeks pre treatment and 10 weeks, 3 months and 12 months post treatment
  Change from baseline in anxiety symptoms. Spence Child Anxiety Scale C/P (SCAS-C/P).

CONTACTS AND LOCATIONS:
Locations (1):
- Barn-och ungdomspsykiatrin, Stockholm, Stockholm, Sweden

REFERENCES:
- [Derived] Vigerland S, Serlachius E, Thulin U, Andersson G, Larsson JO, Ljotsson B. Long-term outcomes and predictors of internet-delivered cognitive behavioral therapy for childhood anxiety disorders. Behav Res Ther. 2017 Mar;90:67-75. doi: 10.1016/j.brat.2016.12.008. Epub 2016 Dec 14. PMID 28012300
- [Derived] Vigerland S, Ljotsson B, Thulin U, Ost LG, Andersson G, Serlachius E. Internet-delivered cognitive behavioural therapy for children with anxiety disorders: A randomised controlled trial. Behav Res Ther. 2016 Jan;76:47-56. doi: 10.1016/j.brat.2015.11.006. Epub 2015 Nov 19. PMID 26649465